CLINICAL TRIAL: NCT00002596
Title: RANDOMIZED MULTIINSTITUTIONAL PHASE III TRIAL OF BEP AND HIGH DOSE CHEMOTHERAPY VERSUS BEP ALONE IN PREVIOUSLY UNTREATED PATIENTS WITH POOR RISK GERM CELL TUMORS
Brief Title: Combination Chemotherapy With or Without Bone Marrow or Stem Cell Transplantation in Treating Men With Untreated Germ Cell Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: SWOG-9442; MSKCC-94076; CLB-99812; E-3894; CDR0000063820 (Registry Identifier: PDQ (Physician Data Query)); NCI-T94-0086D
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2003-10

CONDITIONS: Childhood Germ Cell Tumor; Extragonadal Germ Cell Tumor; Testicular Germ Cell Tumor
Keywords: stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; testicular seminoma; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; extragonadal germ cell tumor; childhood teratoma; childhood malignant testicular germ cell tumor; childhood extragonadal germ cell tumor
MeSH Terms: conditions — Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Carcinoma, Embryonal | interventions — Bleomycin; Filgrastim; Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not known whether combining chemotherapy with bone marrow or peripheral stem cell transplantation is more effective than combination chemotherapy alone in treating men with germ cell tumors.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy with or without bone marrow or peripheral stem cell transplantation in treating men with previously untreated germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of bleomycin, etoposide, and cisplatin (BEP) with or without high-dose carboplatin, etoposide, and cyclophosphamide plus autologous bone marrow or peripheral blood stem cell transplantation in male patients with poor- or intermediate-risk germ cell tumors.
* Compare the toxicity of these regimens in these patients.
* Compare prospectively the prognosis in terms of the rate of decline of the serum tumor markers, human chorionic gonadotropin (hCG) and alpha-fetoprotein (AFP), in patients treated with these regimens.
* Correlate hCG and AFP with complete response and survival in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and risk status (poor vs intermediate). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bleomycin IV on days 1, 8, and 15 and etoposide (VP-16) IV over 30-60 minutes and cisplatin (CDDP) IV over 30-60 minutes on days 1-5 (BEP). Filgrastim (G-CSF) is administered subcutaneously (SC) on days 7-16 or until blood counts recover. Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. G-CSF is discontinued 24 hours before initiating subsequent courses of chemotherapy, and withheld on days of bleomycin administration.
* Arm II: Patients receive 2 courses of BEP and G-CSF as in arm I. Patients who have no marrow involvement with tumor undergo harvest of autologous bone marrow before the first or second course of BEP. Patients who have bone marrow involvement with tumor undergo harvest of G-CSF-mobilized autologous peripheral blood stem cells (PBSC) on days 17-21 of the first and/or second courses of BEP. When blood counts recover, patients receive high-dose intensification comprising carboplatin IV over 1 hour, VP-16 IV over 30-60 minutes, and cyclophosphamide IV over 1 hour on days -5 to -3. Autologous bone marrow or PBSC are reinfused over 15-20 minutes on day 0. G-CSF is administered SC beginning 24 hours after transplantation and continuing until blood counts recover. Beginning 1-3 weeks after hospital discharge for the first transplantation and after recovery from any toxic effects, patients with a Karnofsky performance status of 70-100% receive a second course of high-dose intensification plus a second bone marrow or PBSC transplantation in the absence of disease progression or unacceptable toxicity.

Patients on both arms with brain metastases at presentation undergo radiotherapy and/or surgery concurrently with BEP, if medically indicated.

Patients with normal alpha fetoprotein (AFP) and human chorionic gonadotropin (hCG) tumor marker levels after completion of treatment on arm I or II undergo surgical resection of all residual masses. Patients who have no residual malignant tumor or undergo complete resection of only a mature teratoma receive no further therapy. Patients on arm I who undergo complete resection of residual malignant tumor receive 2 additional courses of VP-16 and CDDP without bleomycin. Patients on arm II who undergo complete resection of residual malignant tumor receive no additional chemotherapy. Patients with an unresectable residual malignant tumor receive additional therapy at the discretion of the treating physician. Patients with residual tumor marker (AFP and hCG) positivity after treatment on arm I or II undergo resection of residual masses if tumor marker values fall to normal by marker half-life.

PROJECTED ACCRUAL: A total of 270 patients (135 per treatment arm) will be accrued for this study within 4.4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven poor-risk, nonseminoma germ cell tumor

  * Must meet 1 of the following 3 conditions:

    * Testis or retroperitoneal primary site without visceral metastasis but with any of the following tumor marker values:

      * Lactic dehydrogenase (LDH) greater than 10 times upper limit of normal (ULN)
      * Human chorionic gonadotropin (hCG) greater than 50,000 IU/L
      * Alpha-fetoprotein (AFP) greater than 10,000 ng/mL
    * Testis or retroperitoneal primary site with 1 or more nonpulmonary visceral metastases (regardless of tumor marker values), including the following:

      * Bone
      * Brain
      * Liver
      * Other nonpulmonary viscera (e.g., skin, spleen)
    * Mediastinal primary site, regardless of presence/absence of visceral metastasis or tumor marker values OR
* Histologically proven intermediate-risk, nonseminoma germ cell tumor

  * Testis or retroperitoneal primary site with no visceral metastasis (except lung), and with any of the following tumor marker values:

    * LDH 3-10 times ULN
    * hCG 5,000-50,000 IU/L
    * AFP 1,000-10,000 ng/mL OR
* Histologically proven intermediate-risk, seminoma germ cell tumor with 1 or more nonpulmonary visceral metastases (regardless of tumor marker values or primary site), including the following:

  * Bone
  * Brain
  * Liver
  * Other nonpulmonary visceral metastasis (e.g., skin, spleen)
* Histologic confirmation may be delayed, at the discretion of the protocol chairman, until after initiation of study therapy for patients with a testicular mass and elevated AFP or hCG if medical circumstances warrant immediate treatment
* Measurable or evaluable disease
* Concurrent registration on protocol MSKCC-89076 (SWOG-9345) for tumor biology studies required

PATIENT CHARACTERISTICS:

Age:

* 12 and over

Sex:

* Male

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* See Disease Characteristics

Renal:

* Creatinine no greater than ULN* OR
* Creatinine clearance greater than 50 mL/min* NOTE: * Abnormal levels due to ureteral obstruction by tumor allowed at the discretion of the protocol chairman

Other:

* HIV negative
* No other concurrent malignancy except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 30 days since prior radiotherapy except for brain metastases or documented disease progression
* Recovered from the toxic effects of any prior radiotherapy

Surgery:

* Recovered from the effects of any recent surgery

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 1994-09; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Patrick J. Loehrer, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center; Kim A. Margolin, MD, Study Chair — City of Hope Comprehensive Cancer Center; Eric J. Small, MD, Study Chair — University of California, San Francisco
Locations (153):
- United States (149):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - St. Joseph Hospital - Orange, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - John Muir Medical Center, Walnut Creek, California
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Hospital Comprehensive Cancer Center, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Helen and Harry Gray Cancer Institute at Good Samaritan Medical Center, West Palm Beach, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Saint Anthony Medical Center, Rockford, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alegent Health-Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - NorthEast Oncology Associates, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Oregon Cancer Institute, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Mary's Medical Center, Huntington, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Ministry Medical Group - Northern Region, Rhinelander, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- Puerto Rico (2):
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Result] Motzer RJ, Nichols CJ, Margolin KA, Bacik J, Richardson PG, Vogelzang NJ, Bajorin DF, Lara PN Jr, Einhorn L, Mazumdar M, Bosl GJ. Phase III randomized trial of conventional-dose chemotherapy with or without high-dose chemotherapy and autologous hematopoietic stem-cell rescue as first-line treatment for patients with poor-prognosis metastatic germ cell tumors. J Clin Oncol. 2007 Jan 20;25(3):247-56. doi: 10.1200/JCO.2005.05.4528. PMID 17235042
- [Result] Bajorin DF, Nichols CR, Margolin KA, et al.: Phase III trial of conventional-dose chemotherapy alone or with high-dose chemotherapy for metastatic germ cell tumors (GCT) patients (PTS): a cooperative group trial by Memorial Sloan-Kettering Cancer Center, ECOG, SWOG, and CALGB. [Abstract] J Clin Oncol 24 (Suppl 18): A-4510, 2006.